CLINICAL TRIAL: NCT05683353
Title: Mechanism and Immune Function Analysis of SARS-CoV-2 Infection in Hematologic Tumors and Discovery of Potential Drug Targets
Brief Title: Mechanism and Immune Function Analysis of SARS-CoV-2 Infection in Hematologic Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yujun DONG, chief of department of hematology, Peking University First Hospital
Other Study IDs: PekingUFH_
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2 Infection; Hematologic Malignancy
Keywords: SARS-CoV-2 infection; hematologic malignancy; leukemia; interaction; immune function; network analysis
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms; Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells are extracted to perform RNA-sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with SARS-CoV-2 positive hematologic tumors: Patients with SARS-CoV-2 positive hematologic tumors over 18 years old excluding patients with severe diseases associated with other systems.
  Interventions: Other: None intervention
- People with SARS-CoV-2 positive without underlying diseases: People with SARS-CoV-2 positive without underlying diseases over 18 years old excluding people with severe diseases associated with other systems.
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention — None intervention.

SUMMARY:
The goal of this observational study is to compare the immune function and infection mechanism of patients with hematologic tumors and those people without underlying diseases after infection with SARS-CoV-2. Clinical characteristics, treatment options and responses will be collected. Peripheral blood will be collected from patients with hematologic tumors infected with SARS-CoV-2 and those people without underlying diseases infected with SARS-CoV-2.

DETAILED DESCRIPTION:
To establish a retrospective and prospective cohort of patients with hematologic tumors infected with SARS-CoV-2 and people without underlying diseases infected with SARS-CoV-2. Firstly, peripheral blood samples will be collected at infection time points and after SARS-CoV-2 nucleic acid testing turns negative. Subsequently, the transcriptome sequencing and immunological experiments will be performed to analyze the differentially expressed genes, immune function of cells, etc.

Comparative analysis:

1. To compare the immune function of patients with hematologic tumors and those without underlying diseases after infection with SARS-CoV-2.
2. The transcriptomic and proteomic changes of patients with hematologic tumors are compared with those without underlying diseases after infection with SARS-CoV-2.
3. From the perspective of complex (human protein interaction subnetwork), the dynamic change process of SARS-CoV-2-targeted human protein complex (periodic complex) was deeply explored, in order to further analyze its potential dynamic infection mechanism and provide new clues for the discovery of drug targets.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of hematologic tumors Clinical diagnosis of SARS-CoV-2 infection

Exclusion Criteria:

- Severe diseases associated with other systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with SARS-CoV-2 positive hematologic tumors over 18 years old.
  People with SARS-CoV-2 positive without underlying diseases over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mechanism and Immune Function Analysis of SARS-CoV-2 Infection in Hematologic Tumors | 1 year
  To compare the infection mechanism and immune function of patients with hematologic tumors infected with SARS-CoV-2 and people infected with SARS-CoV-2 without underlying diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Naranbhai V, Nathan A, Kaseke C, Berrios C, Khatri A, Choi S, Getz MA, Tano-Menka R, Ofoman O, Gayton A, Senjobe F, Zhao Z, St Denis KJ, Lam EC, Carrington M, Garcia-Beltran WF, Balazs AB, Walker BD, Iafrate AJ, Gaiha GD. T cell reactivity to the SARS-CoV-2 Omicron variant is preserved in most but not all individuals. Cell. 2022 Mar 17;185(6):1041-1051.e6. doi: 10.1016/j.cell.2022.01.029. Epub 2022 Feb 3. PMID 35202566
- [Background] Bange EM, Han NA, Wileyto P, Kim JY, Gouma S, Robinson J, Greenplate AR, Hwee MA, Porterfield F, Owoyemi O, Naik K, Zheng C, Galantino M, Weisman AR, Ittner CAG, Kugler EM, Baxter AE, Oniyide O, Agyekum RS, Dunn TG, Jones TK, Giannini HM, Weirick ME, McAllister CM, Babady NE, Kumar A, Widman AJ, DeWolf S, Boutemine SR, Roberts C, Budzik KR, Tollett S, Wright C, Perloff T, Sun L, Mathew D, Giles JR, Oldridge DA, Wu JE, Alanio C, Adamski S, Garfall AL, Vella LA, Kerr SJ, Cohen JV, Oyer RA, Massa R, Maillard IP, Maxwell KN, Reilly JP, Maslak PG, Vonderheide RH, Wolchok JD, Hensley SE, Wherry EJ, Meyer NJ, DeMichele AM, Vardhana SA, Mamtani R, Huang AC. CD8+ T cells contribute to survival in patients with COVID-19 and hematologic cancer. Nat Med. 2021 Jul;27(7):1280-1289. doi: 10.1038/s41591-021-01386-7. Epub 2021 May 20. PMID 34017137
- [Background] Ni L, Ye F, Cheng ML, Feng Y, Deng YQ, Zhao H, Wei P, Ge J, Gou M, Li X, Sun L, Cao T, Wang P, Zhou C, Zhang R, Liang P, Guo H, Wang X, Qin CF, Chen F, Dong C. Detection of SARS-CoV-2-Specific Humoral and Cellular Immunity in COVID-19 Convalescent Individuals. Immunity. 2020 Jun 16;52(6):971-977.e3. doi: 10.1016/j.immuni.2020.04.023. Epub 2020 May 3. PMID 32413330
- [Background] Auwul MR, Rahman MR, Gov E, Shahjaman M, Moni MA. Bioinformatics and machine learning approach identifies potential drug targets and pathways in COVID-19. Brief Bioinform. 2021 Sep 2;22(5):bbab120. doi: 10.1093/bib/bbab120. PMID 33839760
- [Background] Yang S, Fu C, Lian X, Dong X, Zhang Z. Understanding Human-Virus Protein-Protein Interactions Using a Human Protein Complex-Based Analysis Framework. mSystems. 2019 Apr 9;4(2):e00303-18. doi: 10.1128/mSystems.00303-18. eCollection 2019 Mar-Apr. PMID 30984872